CLINICAL TRIAL: NCT02540616
Title: Transcranial Electrical Stimulation for Mal de Debarquement Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study hypothesis was faulty
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-006-01
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Mal de Debarquement Syndrome
Keywords: MdDS; TES; TMS
MeSH Terms: conditions — Mal de debarquement | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a real vs a sham stimulation arm. The sham arm will be offered real treatment after unblinding.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Electrical Stimulation-Real (Experimental): The participant will perform real TES. The forms of TES used in this study will include transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), or transcranial random noise stimulation (tRNS). Each stimulation session will last for 20-minutes.
  Interventions: Device: Transcranial Electrical Stimulation
- Transcranial Electrical Stimulation-Sham (Sham Comparator): The participant will perform sham TES for 20-minutes. The form of sham TES will depend on the active arm, e.g. if tACS is on the active arm, then the sham tACS will be a different frequency of stimulation. If tDCS is the active arm, then a short ramp up of tDCS followed by a ramp down (about 60-seconds) will be used as the sham arm.
  Interventions: Device: Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Transcranial Electrical Stimulation — A form of external neuromodulation using electrodes on the surface of the head. We will be using the TCT tDCS device (www.trans.cranial.com) or devices constructed by our research group or collaborators.
  Other Names: Transcranial Direct Current Stimulation (tDCS); Transcranial Alternating Current Stimulation (tACS); Transcranial Random Noise Stimulation (tRNS); Sham Transcranial Stimulation

SUMMARY:
The goal of this study is to determine whether external neuromodulation using transcranial electrical stimulation (TES) can reduce the perception of self-motion that is experienced by patients with MdDS. Mal de debarquement is translated as the "sickness of disembarkment," and refers to the chronic feeling of rocking dizziness that occurs after exposure to passive motion. A similar form of rocking dizziness can be experienced without a motion trigger in individuals with certain risk factors.

Treatment for MdDS is limited and morbidity is high.The goal of the study is to determine whether TES can suppress the rocking dizziness of MdDS either as a standalone therapy or as an adjunctive therapy to other forms of neuromodulation such as transcranial magnetic stimulation. The investigators will determine the optimal treatment duration and stimulation parameters.

DETAILED DESCRIPTION:
Eligible participants who meet study criteria and pass the safety screen will be invited to participate in the study. If TES is used as add-on treatment to repetitive transcranial magnetic stimulation (rTMS), the training for TES application will be done on-site. However, in a portion of the study that does not involve rTMS, remote training will be performed via a webcam provided that a suitable "Study Buddy" is available to assist the participant.

Participants will maintain web-based diaries of their symptoms for up to four weeks prior to treatment with TES. Before the actual treatment sessions are started, the subjects will complete baseline questionnaires online which will be repeated once a week for up to 12 weeks. Over the course of the study, the subjects will also keep a daily log of their sessions such as how many sessions they performed, for how long, and whether they had any side effects with each session.

The studies will include a sham arm, allocated at a ratio of 1:1. On-site studies will involve the application of EEG, MRI, balance, cognitive, and visual/auditory stimulation tests.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Willing and capable of interacting with the informed consent process
3. Primary disorder being a persistent perception of motion with no other cause determined after a careful interview.
4. Able to identity a study buddy and provide contact information

Exclusion Criteria:

1. Subjects who cannot comply with study conditions.
2. Active psychiatric condition such as mania or psychosis
3. Unstable medical condition
4. Implanted metal in the head or neck (metal or shrapnel, deep brain stimulators, aneurysm clips, cochlear stimulators, retinal implants, etc). Dental fillings are acceptable.
5. Any active skin disorder that affects skin integrity of the scalp.
6. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | 10 years
  This is a well validated 100 point self-reported scale with Functional, Physical, and Emotional components.

SECONDARY OUTCOMES:
Mal de Debarquement Balance Rating Scale | 10 years
  This is a 10 point self-reported scale that assesses the severity of rocking dizziness and its effect on balance function.
Hospital Anxiety and Depression Scale | 10 years
  This is a well validated 42 point self-reported scale of anxiety and dizziness.

OTHER OUTCOMES:
SF-12 | 10 years
  Well established Quality of Life Scale
Motion Sickness Susceptibility Scale | 10 years
  Measures motion sickness susceptibility before and after age 12
Neo-Five Factor Inventory | 10 years
  Quantifies the five major personality traits
Empathy Quotient | 10 years
  40 item online or 20 item abbreviated scale to determine strength of empathic traits
Functional Activities Scale | 10 years
  Measures comfort with doing some basic activities of daily living
Memory Questionnaire | 10 years
  Measures subjective impressions of prospective and retrospective memory
Multidimensional Fatigue Inventory | 10 years
  Measures general, physical, and mental fatigue
Edinburgh Handedness Scale | 10 years
  Standard measure of handedness

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Hee Cha, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be shared once recruitment is sufficient to prevent the inadvertent identification of participants by demographic or clinical characteristics

REFERENCES:
- [Derived] Cha YH, Gleghorn D, Doudican BC. Double-blind randomized N-of-1 trial of transcranial alternating current stimulation for mal de debarquement syndrome. PLoS One. 2022 Feb 4;17(2):e0263558. doi: 10.1371/journal.pone.0263558. eCollection 2022. PMID 35120184